CLINICAL TRIAL: NCT02219646
Title: Monitoring of Endothelial Dysfunction During Chronic Administration of Vardenafil in Patients With Type 2 Diabetes Mellitus: A Longitudinal, Randomised, Placebo-controlled, Double Blind, Phase II b, Clinical Trial
Brief Title: Diabetes & Vardenafil
Acronym: DiVa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda USL Modena (Other)
Responsible Party: Principal Investigator, Manuela Simoni, Ordinary Professor, Azienda USL Modena
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: EudraCT number 2009-014137-25
Record Dates: First submitted 2014-07-24; First posted 2014-08-19 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Endothelial Dysfunction; Erectile Dysfunction
Keywords: T2DM; ED
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vardenafil (Experimental): The study protocol consists of a Screening/Enrolment Phase lasting up to 4 weeks, a Treatment Phase of 24 weeks, and Follow-up/Observation Treatment-free Phase of 24 weeks after the Treatment Phase. During treatment phase, patients enrolled in the Study Group were treated with vardenafil 10 mg twice/daily.
  Interventions: Drug: Vardenafil
- Control (Placebo Comparator): The study protocol consists of a Screening/Enrolment Phase lasting up to 4 weeks, a Treatment Phase of 24 weeks, and Follow-up/Observation Treatment-free Phase of 24 weeks after the Treatment Phase. During treatment phase, patients enrolled in the Control Group were treated with tablets twice/daily identical to the Study Group, but containing placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vardenafil — Vardenafil 10 mg twice daily for six months
  Other Names: Levitra
  Arms: Vardenafil
Drug: Placebo — Placebo two tablets daily for 6 months
  Arms: Control

SUMMARY:
Given the protective effect of nitric oxide (NO) on the endothelium and the results obtained so far in short-term, continuous treatment with phosphodiesterase-5 (PDE5) inhibitors on parameters of endothelial function, we hypothesise that chronic treatment with vardenafil can prevent or delay the deterioration of systemic endothelial function in patients with type 2 diabetes mellitus. The favourable effect of PDE5 inhibitors on sexual function in these patients has been convincingly demonstrated in the past. Here we hypothesise that vardenafil treatment can have beneficial effects on the vascular physiology in other body districts, possibly preventing the development of microangiopathy and atherosclerotic cardiovascular disease in these patients.

The main goal of this study is therefore to monitor the endothelial dysfunction during continuous treatment with vardenafil for 6 months; object of the study will be endothelin 1 and other known parameters of endothelial damage in newly diagnosed patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Phosphodiesterase-5 (PDE5) inhibitors are currently used in the therapy of erectile dysfunction (ED), which is considered to be an early symptom of cardiovascular disease (CD). Impairment of endothelial function is the early lesion preceding atherosclerosis and is common to ED, CD and vascular complications of diabetes mellitus (DM). Continuous administration of the PDE5 inhibitors tadalafil or sildenafil for four weeks in men with increased cardiovascular risk or type 2 DM has been shown to improve endothelial function measured by flow-mediated dilation and reduction of inflammatory markers. The goal of this study is to investigate whether chronic, long-term treatment with vardenafil improves and/or prevents deterioration of systemic endothelial function in patients with type 2 DM. Study design: longitudinal, double-blind, randomised, placebo-controlled interventional study. Patients: 106 male patients (n determined by power analysis) with type 2 DM diagnosed and classified according to the guidelines of the European Association for the Study of Diabetes. Beside the antidiabetic treatment, patients will be randomly assigned to receive either placebo or vardenafil, 10 mg p.o. two times a day for 24 weeks. Exclusion criteria: all contraindications to treatment with PDE5 inhibitors. Age range: 40-60 years. Sample size determined by power analysis assuming variations of the primary end point of ± 10% from baseline at 0.05 α level with a power of 80%, a two-sided test and a dropout rate of 15%. Primary end point: serum endothelin 1 levels (decreased/not increased in the verum group vs. not decrease/increased in the placebo group). Other parameters and measurements: Complete clinical workup, weight, height, waist-hip ratio, serum lipids and glucose, hemoglobin glycated (HbA1c), micro- and macroalbuminuria, homocysteine, high reactive C-protein (hsCRP), interleukin-6 (IL-6), Tumor necrosis factor (TNF)α, fibrinogen, adiponectin, testosterone, sex hormone-binding globulin (SHBG) and estradiol. All parameters measured at baseline, 4 weeks, 12 weeks and 24 weeks on medication as well as 4 and 24 weeks after discontinuation of the study drug. Study duration: two years. Statistics: descriptive statistics, ANCOVA and multiple regression analysis or non-parametric tests as appropriate by STATA. Ethics: The trial will be registered. Ethics committee approval and patient informed consent will be obtained. Expected outcome and objective: Monitoring of endothelial function deterioration in type 2 DM during chronic administration of Vardenafil. Possibility for a long term-follow up study. Publication in a high impact factor journal.

ELIGIBILITY:
Inclusion Criteria:

* Male gender
* Signed written Consent Form
* Type 2 diabetes mellitus diagnosed within 5 years before enrolment in the study
* Body Mass Index (BMI) < 35
* ED (severe, moderate or light according to the International Index of Erectile Function - erectile function domain score < 26 (Rosen et al. 1997))
* Age range: 40-65 years.

Exclusion Criteria:

* Systemic diseases except type 2 diabetes mellitus
* Absence of ED
* Psychiatric disorders
* All contraindications to treatment with PDE5 inhibitors, such as retinitis pigmentosa, non-arteritic anterior ischaemic optic neuropathy, history of coronary artery disease, recent myocardial infarction, unstable angina, systemic arterial hypotension, nitric-oxide donors therapy, severe hepatic and renal failure.

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-03; Primary Completion 2013-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Endothelin-1 | "6 months"
  change in serum endothelin 1 concentration

SECONDARY OUTCOMES:
Flow Mediated Dilation | "baseline"
  Change of flow mediated dilation evaluated by ultrasonography at brachial artery
Flow Mediated dilation (FMD) | "6 months"
  Change of FMD levels
Flow Mediated Dilation | "One year"
  Change of FMD levels

OTHER OUTCOMES:
carotid Intima Media Thickness | "baseline"
  Change of ultrasonographic evaluation of intima-media thickness at both right and left carotid arteries
carotid Intima Media Thickness (IMT) | "6 months"
  Change in IMT levels
carotid Intima Media Thickness | "One year"
  change in IMT levels

CONTACTS AND LOCATIONS:
Overall Officials: Manuela Simoni, MD, PhD, Principal Investigator — Azienda USL Modena
Locations (1):
- Unit of Endocrinology Azienda USL, Modena, Modena, Italy